CLINICAL TRIAL: NCT05847257
Title: Impact of Co Enzyme Q10 as Adjuvant Therapy to Letrozole on Spermiogram and Sex Hormone in Iraqi Infertile Men; A Comparative Study
Brief Title: Impact of Co Enzyme Q10 as Adjuvant Therapy to Letrozole on Spermiogram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Collaborators: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Mohammed Mahmood Mohammed, Clinical associated professor, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023M01
Record Dates: First submitted 2023-04-10; First posted 2023-05-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Male Reproductive Problem; Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: A prospective clinical study. The study initially included 74 patients, on follow-up 7 cases were lost and the final analysis involved 67 cases. These patients were further divided into two groups randomly, group A (29) patients received letrozole 2.5mg twice weekly for 3 months, and group B (38) patients receive letrozole 2.5mg twice a week plus Co Q10 400 mg per day for 3 months.
  Patients with idiopathic Oligo-Astheno-Teratozoospermia (iOAT) syndrome were selected during their visit to the specialized center of infertility/ Nahrain University. Before taking part, each subject provided their written, informed consent. The duration of this study was from December 2021 till October 2022.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Sham Comparator): group A (29) patients received letrozole 2.5mg twice weekly for 3 months
  Interventions: Drug: Letrozole tablets
- Group B (Experimental): Group B (38) patients receive letrozole 2.5mg twice a week plus Co Q10 400 mg per day for 3 months
  Interventions: Drug: Letrozole tablets; Dietary Supplement: Coenzyme Q10 table

INTERVENTIONS:
Drug: Letrozole tablets — letrozole 2.5mg twice weekly for 3 months
Dietary Supplement: Coenzyme Q10 table — Coenzyme Q10 400 mg per day for 3 months
  Arms: Group B

SUMMARY:
Worldwide infertility affects about 15 % of reproductive-age couples. In many cases, infertility can't be treated, new treatment options with promising value were involved in the recent clinical trials.

DETAILED DESCRIPTION:
We will evaluate the impacts of adding coenzyme Q10 to letrozole on spermiogram and sex hormone in men diagnosed with idiopathic oligo/astheno/ teratozoospermia (iOAT) syndrome.

The study will include 67 patients which will be randomly separated into two groups, Group (A) 29 patients will be treated with letrozole 2.5mg tablet orally twice a week, Group (B) 38 patient will be treated with a combination of letrozole 2.5 mg tablet orally twice a week plus Co-Q10 400mg per day, both groups complete treatment for three months. Semen sample, serum FSH, estradiol (E2), and testosterone (T) were analyzed at day one, and at the end of one, two, and three months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients.
2. Aged 18 - 60 years.
3. Confirmed diagnosis with idiopathic Oligo-Astheno-Teratozoospermia (iOAT) syndrome.

Exclusion Criteria:

1. Patients who have been found to have additional infertility causes, such as varicocele or Obstruction of the ejaculatory duct.
2. Those who have had surgery for male factor infertility.
3. Patients with infections such as STD.
4. Patient with renal or liver disease
5. Incomplete patient data

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All male
Enrollment: 74 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The seminal fluid analysis | change in value from baseline to the end of 1st, 2nd and 3rd month for three consecutive months of treatment
  sperm volume/ ml, Sperm concentration/ml, Total sperm count / ml, Progressive Sperm motility (%), Non-progressive Sperm motility (%), Immotile Sperm (%), Normal Sperm morphology (%)

SECONDARY OUTCOMES:
hormone profile | change in value from baseline to the end of 1st, 2nd and 3rd month for three consecutive months of treatment
  concentration of Serum FSH, concentration of Serum estradiol, and concentration of Serum testosterone

CONTACTS AND LOCATIONS:
Locations (1):
- specialized center of infertility/ Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
All participants demographical and clinical characteristics, and outcome of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication of the study

REFERENCES:
- [Derived] Fadhil EB, Mohammed MM, Alkawaz UM. Impact of coenzyme Q10 as an adjuvant therapy to letrozole on spermiogram results and sex hormone levels in Iraqi men with infertility; randomized open label comparative study. F1000Res. 2024 Jun 10;12:1093. doi: 10.12688/f1000research.131985.3. eCollection 2023. PMID 38957201
- See also: Publication — https://f1000research.com/articles/12-1093/v3
- Available data/document: Individual Participant Data Set: 10.5281/zenodo. — https://zenodo.org/records/8191740 — data of impact of coenzyme Q10 as an adjuvant therapy to letrozole on spermiogram results and sex hormone levels in Iraqi men with infertility; randomized open label comparative study